CLINICAL TRIAL: NCT00282971
Title: A Six Month, Open-label Outpatient, Parallel Group Trial Assessing The Impact Of Inhaled Insulin (Exubera(Registered)) On Glycemic Control In Patients With Type 2 Diabetes Mellitus Who Are Poorly Controlled On Two Oral Anti-diabetic Agents
Brief Title: A Clinical Trial Assessing The Impact Of Inhaled Insulin On Glucose Control In Patients With Type 2 Diabetes Mellitus
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Terminated as marketing of this product will be discontinued
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A2171063; EXACTA (Other: Alias Study Number); 2005-003504-11 (EudraCT Number)
Record Dates: First submitted 2006-01-26; First posted 2006-01-27 (Estimated); Results first posted 2009-08-26 (Estimated); Last update posted 2019-04-02 (Actual); Status verified 2019-04

CONDITIONS: Diabetes Mellitus Type 2
Keywords: Type 2 diabetes melllitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Exubera; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Inhaled Insulin (Experimental): Inhaled insulin plus oral therapy
  Interventions: Drug: Inhaled Insulin (Exubera)
- Standard of Care (Other): Standard of Care: All licensed diabetes drugs can be prescribed per discretion of investigators
  Interventions: Other: Standard of Care

INTERVENTIONS:
Drug: Inhaled Insulin (Exubera) — Addition of inhaled insulin to pre-existing oral diabetes therapy.
  Arms: Inhaled Insulin
Other: Standard of Care — Standard of Care: All licensed diabetes drugs can be prescribed per discretion of investigators
  Arms: Standard of Care

SUMMARY:
To assess the impact on glucose control by inhaled insulin in patients with type 2 diabetes who are not well controlled on 2 or more oral anti-diabetic agents

ELIGIBILITY:
Inclusion Criteria:

* Diabetes mellitus type 2
* Failing two or more oral anti-diabetic agents

Exclusion Criteria:

* Asthma, COPD
* Smoking

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 354 (Actual)
Dates: Start 2006-03-06 (Actual); Primary Completion 2008-02-19 (Actual); Study Completion 2008-02-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (64):
- Canada (14):
  - Gain Medical Center, Coquitlam, British Columbia
  - Misericordia Health Centre, Winnipeg, Manitoba
  - Maritime Research Center, Bathurst, New Brunswick
  - Office of Dr. Salim Sunderji, London, Ontario
  - Orillia Soldier's Memorial Hospital, Orillia, Ontario
  - Douglas Tweel M.D. Professional Corporation, Charlottetown, Prince Edward Island
  - Laboratoire Sante Le Gaspesien Inc., Bonaventure, Quebec
  - Centre de santé et de services sociaux de Chicoutimi, Centre de médecine genique communataire, Chicoutimi, Quebec
  - Rhodin Recherche Clinique, Drummondville, Quebec
  - Q & T Research Outaouais Inc., Gatineau, Quebec
  - Hopital Charles LeMoyne, Greenfield Park, Quebec
  - Hopital Laval, Saint-Foy, Quebec
  - Centre Medical des Carrieres, Saint-Marc-des-Carrieres, Quebec
  - CIC Mauricie Inc., Trois-Rivières, Quebec
- France (16):
  - Hotel Dieu CHU, Clinique d´Endocrinologie, Maladie Metaboliques, Nutrition, Nantes, Cedex 01
  - Groupe Hospitalier Sud/Service d'Endocrinologie, Amiens
  - Private Practise, Armentières
  - Service d'Endocrinologie-, Bondy
  - Hopital LA Cavale Blanche, Service de Diabetologie, Brest
  - CHU Cote de Nacre, Service d'Endocrinologie, Cean Cedex
  - Private Practise, Chartres
  - Office of Antoine Lemaire, MD, Lille
  - Centre Hospitalier Bretagne Sud, Lorient
  - Hopital Lapeyronnie Sce des Maladies, Montpellier
  - Hopital Saint Michel, Paris
  - Hopital Bichat, Service d'Endocrinology, Paris
  - Hopital Robert Debre, Reims
  - C.H. Sud, Diabetologie, Rennes
  - Centre Hospitalier Victor Provo, Roubaix
  - Hôpital Jeanne d'Arc - Dommartin les Toul, Toul
- Greece (5):
  - General Hospital of Athens "Laikon", 1st Propedeutic University Internal Medicine Clinic, Athens
  - "Hygeia" Diagnostic and Therapeutic Center of Athens, Diabetes Clinic, Athens
  - "ATTIKON" University General Hospital, 2nd Propedeutic University Internal Medicine Clinic, Haidari
  - Peripheral General Hospital of Nikaia "Ag. Panteleimon", Internal Medicine Department, Pireaus
  - University General Hospital of Thessaloniki "A.H.E.P.A." 1st Propedeutic University Internal Medicin, Thessaloniki
- Portugal (6):
  - Hospital Infante D. Pedro, Aveiro
  - Hospitais da Universidade de Coimbra, Coimbra
  - Associação Protectora dos Diabéticos de Portugal, Lisbon
  - Serviço de Endocrinologia - Hospital de Egas Moniz, Lisbon
  - Hospital Geral de Santo António, Porto
  - Centro Hospitalar de Torres Vedras, Torres Vedras
- Spain (17):
  - Hospital Clinico Universitario de Santiago, Santiago de Compostela, A Coruña
  - Hospital de Conxo, Santiago de Compostela, A Coruña
  - Hospital de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital Mutua de Terrassa, Terrassa, Barcelona
  - Clinica Universitaria de Navarra, Pamplona, Navarre
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Hospital General Universitario de Alicante, Alicante
  - Hospital de La Santa Creu I Sant Pau, Barcelona
  - Hospital General Universitario Valle de Hebron, Barcelona
  - Hospital Universitario Puerta de Hierro, Madrid
  - Hospital 12 de Octubre, Madrid
  - Hospital de Mostoles, Madrid
  - Complejo Hospitalario Carlos Haya Hospital Civil - Pabellon C, Málaga
  - Hospital Montecelo, Pontevedra
  - Hospital Universitario La Fe, Valencia
  - Hospital Clinico Universitario de Valencia, Valencia
  - Hospital Clinico Universitario Lozano Blesa, Zaragoza
- Sweden (3):
  - Ängelholms sjukhus, Ängelholm
  - Sodersjukhuset, Stockholm
  - Karolinska US Huddinge, Stockholm
- Turkey (Türkiye) (3):
  - Hacettepe University Medical School Department of Endocrinology, Ankara
  - Istanbul University Istanbul Medical School, Department of Endocrinology, Istanbul
  - Dokuz Eylul University Medical School, Department of Endocrinology, Izmir

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A2171063&StudyName=A%20Clinical%20Trial%20Assessing%20The%20Impact%20Of%20Inhaled%20Insulin%20On%20Glucose%20Control%20In%20Patients%20With%20Type%202%20Diabetes%20Mellitus

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Total subjects enrolled=354. Total subjects given study drug=351. (ie, 3 subjects withdrew after enrollment/randomization, but prior to receiving study drug)
Period: Overall Study
Arm/Group | Inhaled Insulin | Standard of Care
Started | 180 | 171
Completed | 146 | 149
Not Completed | 34 | 22

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Inhaled Insulin | Standard of Care | Total
Number analyzed (Participants) | 180 | 171 | 351
Age, Customized [Number; unit: participants]
  <18 years | 0 | 0 | 0
  Between 18 and 44 years | 12 | 6 | 18
  Between 45 and 64 years | 112 | 113 | 225
  >=65 years | 56 | 52 | 108
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76 | 80 | 156
  Male | 104 | 91 | 195

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change From Baseline in Glycosylated Hemoglobin (HbA1c) at Week 24
Description: [(week 24 value - baseline value)/baseline value]*100%
Time Frame: 4, 12 and 24 weeks
Population: Out of 180 and 171 subjects that were treated with study drug and usual care, respectively, the Full Analysis Set (FAS)for each group which was analyzed for efficacy, was 179 and 170 subjects, respectively.
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Inhaled Insulin | Standard of Care
Number analyzed (Participants) | 179 | 170
percentage change
  week 4 (n=164 and 158, respectively) | -1.08 (0.61) | -0.62 (0.55)
  week 12 (n=159 and 150, respectively) | -2.03 (0.97) | -1.37 (0.92)
  week 24 (n=142 and 150, respectively) | -2.02 (1.10) | -1.44 (1.10)
  week 24 (LOCF, n=175 and 170, respectively) | -1.94 (1.09) | -1.42 (1.09)

2. Secondary Outcome: Percentage of Participants Achieving Glycemic Control by Visit
Description: 2 definitions of good glycemic control were used: an HbA1c result of ≤6.5% or ≤7.0%
Time Frame: 4, 12 and 24 weeks
Population: Out of 180 and 171 subjects that were treated with study drug and usual care, respectively, the Full Analysis Set (FAS)for each group which was analyzed for efficacy, was 179 and 170 subjects, respectively. LOCF=last observation carried forward.
Measure: Number; unit: Percentage of participants
Arm/Group | Inhaled Insulin | Standard of Care
Number analyzed (Participants) | 179 | 170
Percentage of participants
  HbA1c<=7% at week 4 (n=165 and 158 respectively) | 6.1 | 0.0
  HbA1c<=7% at week 12 (n=160 and 150 respectively) | 38.1 | 11.3
  HbA1c<=7% at week 24 (n=143 and 150 respectively) | 34.3 | 12.0
  HbA1c<=7% at wk-24 LOCF (n=178 & 170 respectively) | 32.0 | 12.9
  HbA1c<=6.5% at week 4 (n=165 and 158 respectively) | 0.6 | 0.0
  HbA1c<=6.5% at week 12 (n=160 &150 respectively) | 15.6 | 4.7
  HbA1c<=6.5% at week 24 (n=143 &150 respectively) | 18.2 | 6.0
  HbA1c<=6.5% at wk-24 LOCF(n=178 &170 respectively) | 15.2 | 5.9

3. Secondary Outcome: Change From Baseline in FEV1 at Week 24 LOCF
Time Frame: 24 weeks
Population: Out of 180 and 171 subjects that were treated with study drug and usual care, respectively, the Full Analysis Set (FAS)for each group which was analyzed for efficacy, was 179 and 170 subjects, respectively.FEV1=forced expiratory volume in 1 second;LOCF=last observation carried forward.
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | Inhaled Insulin | Standard of Care
Number analyzed (Participants) | 179 | 170
Liter | -0.27 (9.85) | -0.08 (0.61)

ADVERSE EVENTS:
Arm/Group | Inhaled Insulin | Standard of Care
Serious Adverse Events (participants affected / at risk) | 8/180 | 6/171
Other Adverse Events (participants affected / at risk) | 123/180 | 98/171
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Inhaled Insulin (N=180) | Standard of Care (N=171)
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1
Oedema peripheral (General disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Incision site cellulitis (Infections and infestations) | 1 | 0
Device malfunction (Injury, poisoning and procedural complications) | 1 | 0
Blood glucose increase (Investigations) | 1 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Inhaled Insulin (N=180) | Standard of Care (N=171)
Abdominal pain (Gastrointestinal disorders) | 2 | 4
Diarrhoea (Gastrointestinal disorders) | 4 | 3
Asthenia (General disorders) | 5 | 6
Fatigue (General disorders) | 4 | 3
Pyrexia (General disorders) | 4 | 1
Bronchitis (Infections and infestations) | 5 | 2
Influenza (Infections and infestations) | 6 | 7
Nasopharyngitis (Infections and infestations) | 8 | 4
Upper respiratory tract infection (Infections and infestations) | 5 | 5
Urinary tract infection (Infections and infestations) | 7 | 6
Hypoglycaemia (Metabolism and nutrition disorders) | 118 | 98
Dizziness (Nervous system disorders) | 6 | 3
Headache (Nervous system disorders) | 2 | 6
Tremor (Nervous system disorders) | 8 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 10 | 2
Hypertension (Vascular disorders) | 2 | 4

LIMITATIONS AND CAVEATS:
Study terminated prematurely since the sponsor stopped marketing and manufacturing of EXUBERA and withdrew Market Authorization in Europe in September 2008. No efficacy, safety, or quality reason was associated with the premature halt of this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of <60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), <12 mo from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential info other than study results.